CLINICAL TRIAL: NCT05786118
Title: The Effects of Sacroiliac Joint Dysfunction on Gait and Disability in Patients With Chronic
Brief Title: The Effects of Sacroiliac Joint Dysfunction on Gait and Disability
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Director, Kutahya Health Sciences University
Other Study IDs: CLBP and SIJ
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low-back Pain; Sacroiliac Joint Dysfunction; Gait, Unsteady; Disability Physical
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIJ Group: Individuals with sacroiliac joint dysfunction: Participants will be grouped as positive sacroiliac joint dysfunction according to Laslett's algorithm using provocation tests to detect sacroiliac joint dysfunction.
  Interventions: Other: No intervention
- Control Group: Individuals with no sacroiliac joint dysfunction: Individuals with sacroiliac joint dysfunction: Participants will be grouped as negative sacroiliac joint dysfunction according to Laslett's algorithm using provocation tests to detect sacroiliac joint dysfunction.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study

SUMMARY:
It has been reported that gait coordination changes in patients with chronic low back pain, walking slower, taking shorter steps and having asymmetrical stride lengths compared to their healthy peers. In addition to many factor cause gait dysfunction, sacroiliac joint dysfunction might be one of reason of these problems. A study examining the effects of sacroiliac joint dysfunction on gait and disability in individuals with chronic low back pain has not been found in the literature. Therefore, the aim of this study is to evaluate the gait parameters and disability of individuals with chronic low back pain and to reveal their relationship with sacroiliac joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study.
* Patients with 18-65 years
* Low back pain for at least 3 months,
* Reported pain severity of 2 or greater according to the numeric pain rating scale

Exclusion Criteria:

* Previous spine or lower extremity surgery
* Pregnancy
* Severe hypermobility syndromes
* Severe osteoporosis
* Spondyloarthropathies
* Spondylolisthesis
* Systemic inflammatory diseases
* Any neurological disorder that affects balance and gait

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who directly presented to the Physical Therapy Department of Kutahya Health Sciences University Hospital during the study period with persistent low back pain, will be screened for eligibility by an independent physician (H.H.G.)
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Gate speed of time-distance gait parameters | 1 minutes
  Gate speed will be evaluated using with gait platform. The software gives the outcome as km/h.
Step length of time-distance gait parameters | 1 minutes
  Step lengt will be evaluated using with gait platform. The software gives the outcome as cm and calcules for each lower extremity.
Stride length of time-distance gait parameters | 1 minutes
  Stride length will be evaluated using with gait platform.The software gives the outcome as cm.
Step time of time-distance gait parameters | 1 minutes
  Step time will be evaluated using with gait platform.The software gives the outcome as sec and calcules for each lower extremity.
Stride time of time-distance gait parameters | 1 minutes
  Stride time will be evaluated using with gait platform.The software gives the outcome as sec and calcules for each lower extremity.
Cadance of time-distance gait parameters | 1 minutes
  Cadance time will be evaluated using with gait platform.The software gives the outcome as steps/min.
Center of Pressure path length of balance parameters | 2 minutes
  Center of Pressure path length will be evaluated using with gait platform. The software gives the outcome as mm.
Ellipse area of balance parameters | 1 minutes
  Ellipse area will be evaluated using with gait platform. The software gives the outcome as mm2.

SECONDARY OUTCOMES:
Oswestry Disability Index | 5 minutes
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten questions. Each question is scored on a scale of 0-5. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Numeric Pain Rating Scale | 1 minutes
  The Numeric Pain Rating Scale (NPRS) that is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Ismail S [isaracoglu], P.hD., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University Evliya Celebi Hospital Physical Therapy and Rehabilitation Department, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No